CLINICAL TRIAL: NCT03226730
Title: Evaluating Household Visits and Small Groups to Increase Contraception Use Among Married Adolescent Girls in Rural Niger
Acronym: IMPACT-RMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Pathfinder International (Industry)
Responsible Party: Principal Investigator, Jay G. Silverman, PhD, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 2016-1430
Record Dates: First submitted 2016-10-07; First posted 2017-07-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Contraception
Keywords: Female Adolescent; Married; West Africa; Family Planning; Contraceptive Use; Birth Spacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Household Visits (Experimental): Arm 1 will receive gender synchronized household visits (i.e., visits by a female community health worker to the participating married adolescent female and visits by a male community health worker to the participating husband of the married adolescent female). Approximately 10-12 visits with wives and 4-6 visits with husbands are expected to take place over the course of the project. Study Arms 1-3 will additionally receive community enabling environment activities and adolescent-specific service delivery activities to support adolescent contraception use. Community enabling environment activities will include engaging religious leaders, community leaders, and familial gatekeepers of the married adolescent wives, such as in-laws, in community dialogues on a monthly basis.
  Interventions: Behavioral: Household Visits
- Arm 2: Small Groups (Experimental): This arm will receive, in addition to the community-level components, gender synchronized group-based interventions (i.e., separate group-based interventions for husbands of adolescent wives and adolescent wives, themselves). Male-only and female-only small groups for participating husbands and wives will be held separately on bimonthly and monthly intervals, respectively. In this project, each small group will consist of 10-15 participants and will be held in places participants have deemed safe spaces (e.g., a place that has auditory and visual privacy, is safe for girls to walk to, has been designated by community leaders as a protected place for girls to meet). Approximately 8-10 female small groups and 4-6 male groups are expected to take place over the course of the project.
  Interventions: Behavioral: Small Groups
- Arm 3: Household Visits + Small Groups (Experimental): In addition to the community enabling environment components, this arm will receive a combination of household visit and small groups intervention components, as described above for Arms 1 and 2, in order to understand the combined effect of these two interventions on the outcomes of interest.
  Interventions: Behavioral: Household Visits; Behavioral: Small Groups
- Arm 4: Control (No Intervention): The fourth arm will serve as the control condition. Individuals in these villages will not receive the household, small group, or community-enabling environment intervention components.

INTERVENTIONS:
Behavioral: Household Visits — Household visits will be conducted to build trust in the health system, educate regarding different forms of modern contraception, (how administered, how they work, availability), dispel related myths (i.e., those regarding infertility), promote the health advantages of birth spacing, and create related dialogue among adolescent wives and other household members present during these visits. The relais will provide and resupply oral contraceptive pills and condoms to interested participants and will accompany the married adolescent to the nearest health facility for other forms of contraception, if requested to do so. To complement the household visits to married female adolescents, male relais will conduct home visits to discuss healthy timing and spacing of pregnancy with husbands of adolescent females, provide education on different forms of contraception, and discuss concerns husbands may have regarding use of contraception.
  Arms: Arm 1: Household Visits; Arm 3: Household Visits + Small Groups
Behavioral: Small Groups — In the wife-only groups, adolescent wives will be convened by trained adult female community members to learn and discuss a broad range of gender and health-related topics, with a focus on modern contraception, and cultivate self-efficacy, social support and life skills. The small groups will be led by trained female small group mentors who are trained peers and will follow a designated curriculum consisting of different topics each week developed by Pathfinder International and derived from Population Council/UNFPA's Safe Spaces curriculum. The husband groups will follow a curriculum adapted from Promundo's Program P6 and supplemented by the tools and activities developed by Pathfinder International. These groups of husbands will focus on fostering reflection and dialogue to contribute to more equitable gender norms, support for contraception use for HTSP, positive health seeking behavior for them and their families, and increased couples communication and joint SRH decision-making.
  Arms: Arm 2: Small Groups; Arm 3: Household Visits + Small Groups

SUMMARY:
This study entails a quasi-experimental, mixed-methods (i.e., complementary quantitative and qualitative) outcome evaluation to assess the efficacy of the Reaching Married Adolescents (RMA) Interventions developed and implemented by Pathfinder International to increase contraception use and contraception use intentions among married adolescent girls ages 13-19 in three rural districts of the Dosso region of Niger. Intervention models (gender-synchronized household visits and small groups) will be tested using a randomized 4-arm outcome evaluation design; Arm 1 will receive household visits, Arm 2 will receive small groups; Arm 3 will receive household visits plus small groups, and Arm 4 will serve as the control group and will not receive any intervention. The quantitative component will consist of collecting quantitative baseline, 16-months follow-up, and 27-months survey data from randomly selected married adolescent girls (n=1200) and their husbands (n=1200) who are participating in each Arm of the study. Qualitative elements will include ethnography at two time points and semi-structured in-depth interviews half way through intervention implementation. A costing and cost effectiveness analysis will also be conducted to evaluate which intervention provides the largest gain in the primary outcomes for each dollar spent.

DETAILED DESCRIPTION:
This study entails a quasi-experimental, mixed-methods (i.e., complementary quantitative and qualitative) outcome evaluation to assess the efficacy of the Reaching Married Adolescents (RMA) Interventions to increase contraception use and contraception use intentions among married adolescent girls ages 13-19 in three rural districts of the Dosso region of Niger. Two intervention models (gender-synchronized household visits and small groups) will be tested using a randomized 4-arm outcome evaluation design; Arm 1 will receive household visits, Arm 2 will receive small groups; Arm 3 will receive household visits plus small groups, and Arm 4 will serve as the control group and will not receive any intervention. The quantitative component will consist of collecting quantitative baseline and 16-months follow-up survey data from randomly selected married adolescent girls (n=1200) and their husbands (n=1200) who are participating in each Arm of the study. Qualitative elements will include ethnography at two time points and semi-structured in-depth interviews half way through intervention implementation. A costing and cost effectiveness analysis will also be conducted to evaluate which intervention provides the largest gain in the primary outcomes for each dollar spent.

Quasi-Experimental Quantitative Evaluation Design. The 4-arm RMA outcome evaluation will take place across 48 villages clustered within the 3 districts (i.e., 16 villages per district) in the Dosso region of Niger; specifically, Loga, Doutchi and Dosso. Each of the 3 districts will be assigned to 1 of the 3 intervention conditions. Within each district, 16 comparable villages (i.e., rural, Hausa or Zarma-speaking, at least 1000 inhabitants, similar wealth distribution profile, and located within the specified range of distance from health facilities providing effective contraception) will be randomly selected to be assigned to either the district-specific intervention arm or to the control condition. A stratified randomization approach will be used, in which villages will be stratified into two groups based on the village having or not having a health center co-located in their village. Specifically, within each district, 8 villages will be randomly selected among those that have a co-located health center, and 8 villages will be randomly selected from among those villages that do not have a co-located health center (all within the parameters listed above). Within each of these 2 groupings of 8 villages, 2 villages will be randomly selected to be assigned to the control arm. Thus, 12 villages will be assigned to the intervention and 4 will be assigned to serve as control villages in each district. Each village will act as a cluster, with the unit of analysis being the married female adolescent (ages 13-19 years).

Qualitative Evaluation Design. This evaluation study will employ qualitative methods to complement the proposed quantitative evaluation design. The first method employed will be ethnography (i.e., participant observation, in-depth interviewing, informal discussions) to explore the processes related to changing understanding, intentions and behaviors related to use of modern contraception in the context of participating in the RMA interventions. Three villages in Arm 3 receiving the full complement of the RMA programs (i.e., male and female household visits, and male and female groups) will be the source for ethnographic observational field notes, informal group discussion field notes, and informal interview field notes. Three pairs of trained, local research assistants (6 total; 2 per village) will live with families of adolescent wife participants who are living in three separate villages and will participate in the daily life of the families and broader community (cooking, cleaning, farming, etc.) for a period of two month total, one month corresponding with 3 months and 14 months after program initiation. Research assistants will observe but not participate in household visit and small group interventions. Additionally, they will conduct informal, open-ended interviews and consultations with key respondents throughout the community (male and female RMA participants, older adults including in-laws, local political, business and religious leaders).

Findings of the ethnographic phase will inform a semi-structured interview phase to capture narratives regarding intervention acceptability and the roles of the RMA program in increased knowledge, altered intention and changed behaviors regarding decisions on use of modern contraception, inclusive of a focus on issues of gender equity and persistent barriers to contraception acceptance and use. Forty-eight adolescent wives and husbands of adolescent wives participating in the RMA program, and key informants (e.g., village leaders, health providers, etc.) from intervention Arms 1 and 2 will provide semi-structured interview data (n=24 interviews per study arm). Semi-structured interviews (60 minutes) will be conducted approximately 8 months after implementation is initiated. These data will, in turn, inform the foci of the second round of ethnography to be collected at 14 months post program initiation.

Costing and cost-effectiveness will be calculated for each study arm. If one or more intervention arms are found to be effective at increasing contraception use or intention to use contraception, the investigators will compare the cost effectiveness of achieving the outcomes using the WHO-CHOICE methodology.

The study will take place over the course of 4 years total; rolling recruitment and baseline data collection will take place over a period of 3 months, the intervention will be implemented across 16 months with a rolling start and finish, follow-up (27 months) and endline (45 months) data collection will take place over 3 months. Qualitative ethnography data collection will take place at two time periods; at 3 months and 14 months after intervention implementation begins, one month at each time point. Semi-structured interviews will be conducted approximately half-way between the beginning and end of the intervention implementation, in month 8.

ELIGIBILITY:
Inclusion Criteria:

For Women:

* Married
* 13-19 years old
* Fluent in Hausa or Zarma
* Residing in the village where recruitment is taking place with no plans to move away in next 18 months or plan to travel for more than 6 months during that period
* Providing informed consent.

For Men:

* Must be the husband to an eligible adolescent participating in the study
* Hausa or Zarma speaking
* Providing informed consent.

Exclusion Criteria:

For Women:

* Plans to move away in next 18 months or plans to travel for more than 6 months during that period;
* Currently sterilized (to enable measurement of changes in use of temporary methods of contraception from baseline to 16-months follow-up)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2898 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Contraception Use Questionnaire | baseline and 18 month follow up
  Change in use of effective methods of contraception (methods assessed individually)
Intentions to Use Contraception Questionnaire | baseline and 18 month follow up
  Change in behavioral intentions regarding effective contraceptive use (next 3 months)

SECONDARY OUTCOMES:
Social norms regarding gender equity Questionnaire | baseline and 18 month follow up
  Change in social norms regarding husband physical and sexual violence toward wives, women's autonomy and husband control related to family life
Female Empowerment Questionnaire | baseline and 18 month follow up
  Change in autonomy, decision-making, freedom from violence and control, especially with regard to contraceptive use
Knowledge of effective contraceptive methods Questionnaire | baseline and 18 month follow up
  Change in knowledge of effective contraceptive methods, mechanisms, and common side effects
Acceptance of effective contraceptive methods Questionnaire | baseline and 18 month follow up
  Change in attitudes and beliefs regarding use of contraceptive methods for birth spacing

CONTACTS AND LOCATIONS:
Overall Officials: Jay G Silverman, PhD, Principal Investigator — Center on Gender Equity and Health, University of California, San Diego
Locations (2):
- Center on Gender Equity and Health, University of California, San Diego, San Diego, California, United States
- Pathfinder International, Niamey, Niger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silverman JG, Brooks MI, Aliou S, Johns NE, Challa S, Nouhou AM, Tomar S, Baker H, Boyce SC, McDougal L, DeLong S, Raj A. Effects of the reaching married adolescents program on modern contraceptive use and intimate partner violence: results of a cluster randomized controlled trial among married adolescent girls and their husbands in Dosso, Niger. Reprod Health. 2023 Jun 5;20(1):83. doi: 10.1186/s12978-023-01609-9. PMID 37277837
- [Derived] Challa S, DeLong SM, Carter N, Johns N, Shakya H, Boyce SC, Vera-Monroy R, Aliou S, Ibrahima FA, Brooks MI, Corneliess C, Moodie C, Nouhou AM, Souley I, Raj A, Silverman JG. Protocol for cluster randomized evaluation of reaching married adolescents - a gender-synchronized intervention to increase modern contraceptive use among married adolescent girls and young women and their husbands in Niger. Reprod Health. 2019 Dec 18;16(1):180. doi: 10.1186/s12978-019-0841-3. PMID 31852538